CLINICAL TRIAL: NCT00445471
Title: A Prospective Study Comparing the Mifne Approach of Treating Childhood Autism With Routine Standard Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Mifne began treating younger patients who could not be diagnosed with the ADOS used in the study
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, alan apter, Director, Feinberg Child Study Center and Department of Psychiatry, Schneider's Children's Medical Center of Israel, Rabin Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4222
Record Dates: First submitted 2007-03-08; First posted 2007-03-09 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Child Development Disorders, Pervasive
Keywords: Autism Spectrum Disorder; Autistic Disorder; Pervasive Developmental Disorder
MeSH Terms: conditions — Child Development Disorders, Pervasive; Autism Spectrum Disorder; Autistic Disorder | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): Mifne Approach to PDD
  Interventions: Behavioral: Mifne Approach to PDD
- B (Other): Treatment as usual
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Mifne Approach to PDD
  Arms: A
Behavioral: Treatment as usual
  Arms: B

SUMMARY:
The current study aims at comparing outcomes achieved using the Mifne approach of treating autistic children with results obtained when routine standard treatment is used. A prospective comparative study will be performed comparing the results of 12 children treated at Mifne with 12 children treated with treatment as usual. A child and adolescent psychiatrist using the Autism Diagnostic Interview-Revised (ADI-R) and the Autism Diagnostic Observation Schedule-Generic (ADOS-G) will make the diagnostic assessment and a developmental psychologist will make the developmental and psychological assessments using the Vineland Adaptive Behavior Scales-Revised and the Bayley Scales of Infant Development (BSID II) before the child enters the study. Each child will be reassessed following completion of the Mifne intervention, at three and at six months after commencement of treatment. The control child will also be reassessed at three and at six months after commencement of a therapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:

* All children between the ages of 2-5 years who meet diagnostic criteria for Autism or Pervasive Developmental Disorder by DSM IV criteria who are referred for treatment at Mifne for the treatment group.
* The control group will consist of children meeting the same criteria who are referred to Schneider Children's Medical Center of Israel (SCMCI). Matching will be for age, sex, ethnicity, socioeconomic status, IQ, language development and diagnosis.

Exclusion criteria:

* All referred children who do not meet criteria for Autism or PDD or do not understand Hebrew.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2007-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
ADOS scores at 3 and 6 months after commencement of treatment | 2.5 years

SECONDARY OUTCOMES:
CGI-I score after 3 and 6 months | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Alan Apter, MD, Principal Investigator — Director Department of Psychological Medicine Schneider Children's Medical Center of Israel
Locations (1):
- Schneider Children's Medical Center of Israel, Departemnt of Psychological Medicine, Petah Tikva, Israel